CLINICAL TRIAL: NCT01235637
Title: Efficacy of Alfentanyl Versus Sufentanyl in Children for Pain During Treatment by Tracheal Suction in an Intensive Care Unit.
Brief Title: Alfentanil Versus Sufentanil for Pain in Children During for Tracheal Suction
Acronym: DOLOREAPEDIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCIC 10 10
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Child Comfort; Morphine; Intensive Care Units; Pediatric
Keywords: COMFORT B score; Bis score
MeSH Terms: interventions — Alfentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alfentanil (Active Comparator)
  Interventions: Drug: Alfentanil
- Sufentanil (Sham Comparator)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Alfentanil — dosage form: injectable drug, opioid analgesic morphine, intravenous drug.
  Dosage: 10μg/Kg, dilution: 1 ml = volume equivalent to 66μg or 10μg/kg = 1.43μg/kg fentanyl.
  Frequency and duration: 2 bolus injection before 2 tracheal suctions at 0 and 4 hours respectively.
  Arms: Alfentanil
Drug: Sufentanil — dosage form: injectable drug, opioid analgesic morphine, intravenous drug.
  Dosage: intravenous drug to 0,15 µg/Kg : Blisters of 10 ml, box of 20. MERCK
  Frequency and duration: 2 bolus injection before 2 tracheal suctions at 0 and 4 hours respectively.
  Arms: Sufentanil

SUMMARY:
The main objective is to assess the efficacy of Alfentanil for pain in children treated by tracheal suction in pediatric intensive care units in France, compared to Sufentanyl, the current standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* child between 1 month and 15 years of age
* affiliation to the French social security system or equivalent
* child receiving mechanical ventilation for at least 4 hours and less than 48 hours
* ventilation to be provided for at least 8 hours
* less than 30 days in pediatric intensive care
* child under intravenous sedation
* consent of both parents
* consent of child when possible

Exclusion Criteria:

* curarized child
* ketamine treatment
* children suffering from facial and/or severe brain traumatism
* known hypersensitivity reaction to morphine or intolerance insufficiency to sufentanyl
* respiratory
* chronic obstructive pulmonary disease
* myasthenia
* treatment with morphine agonists-antagonists, or combination with MAOIs
* renal or liver disorders
* preterm birth of more than one month of life (but not at full term by corrected age)
* associated treatment or pathology contra-indicating administration of Sufentanyl epidural

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
COMFORT score | 8 hours
  pain score recommended in pediatric intensive care units in France

SECONDARY OUTCOMES:
Hemodynamic criteria | 8 hours
  blood pressure and heart rate
Bispectral Index score | 8 hours
  assess the level of child's sedation

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle WROBLEWSKI, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Stanik-Hutt JA, Soeken KL, Belcher AE, Fontaine DK, Gift AG. Pain experiences of traumatically injured patients in a critical care setting. Am J Crit Care. 2001 Jul;10(4):252-9. PMID 11432213
- [Background] Ista E, van Dijk M, Tibboel D, de Hoog M. Assessment of sedation levels in pediatric intensive care patients can be improved by using the COMFORT "behavior" scale. Pediatr Crit Care Med. 2005 Jan;6(1):58-63. doi: 10.1097/01.PCC.0000149318.40279.1A. PMID 15636661
- [Background] Triltsch AE, Nestmann G, Orawa H, Moshirzadeh M, Sander M, Grosse J, Genahr A, Konertz W, Spies CD. Bispectral index versus COMFORT score to determine the level of sedation in paediatric intensive care unit patients: a prospective study. Crit Care. 2005 Feb;9(1):R9-17. doi: 10.1186/cc2977. Epub 2004 Nov 10. PMID 15693968
- [Background] Brocas E, Dupont H, Paugam-Burtz C, Servin F, Mantz J, Desmonts JM. Bispectral index variations during tracheal suction in mechanically ventilated critically ill patients: effect of an alfentanil bolus. Intensive Care Med. 2002 Feb;28(2):211-3. doi: 10.1007/s00134-001-1189-y. Epub 2002 Jan 12. PMID 11907667
- [Background] Veyckemans F. [Sedation in children: how and for who?]. Arch Pediatr. 2006 Jun;13(6):835-7. doi: 10.1016/j.arcped.2006.03.131. Epub 2006 May 12. No abstract available. French. PMID 16697580